CLINICAL TRIAL: NCT03255681
Title: Efficacy of Platelet-Rich Plasma Filler for Treatment of Tear Trough Deformities
Brief Title: PRP Administration in the Nasojugal Folds
Acronym: PRP
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: USAF Regulatory Concerns
Sponsor: David Grant U.S. Air Force Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FDG20170008H
Record Dates: First submitted 2017-08-17; First posted 2017-08-21 (Actual); Last update posted 2019-01-04 (Actual); Status verified 2019-01

CONDITIONS: Facial Injuries and Disorders
Keywords: Cosmetics; Filler
MeSH Terms: conditions — Facial Injuries; Disease

STUDY DESIGN:
Intervention Model Description: The study treatment group will have one half of their face treated with PRP filler and the other half of the face treated with PRP with CaCl2. Using a VectraH1 3D camera, the degree of volume achieved, measured in cm3 using VECTRA Capture Analysis module software, will be assessed at one, three and six and twelve month intervals and compared to the pre-procedure imaging. This is therefore a pilot study and results will need to be reviewed after performing this protocol on 50 subjects.
Masking Description: No masking.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Split face study (Experimental): Split face study with the left side of the face receiving PRP injections and the right side of the face receiving PRP with 0.1cc of 10% calcium chloride per 1mL of PRP. The volume of PRP will be used upon the discretion of the provider for treatment of the cosmetic facial deformity but will be in equal amounts for each side on every patient participating in the study.
  Interventions: Procedure: PRP injections into nasojugal folds

INTERVENTIONS:
Procedure: PRP injections into nasojugal folds — A topical anesthetic consisting of 4% Lidocaine (Topicaine) will be placed in the treatment zone prior to injections for no less than 20 minutes per manufactures recommendations.
  11ml of whole blood will be drawn from the patient via venous aspiration into the Eclipse collection tube. The blood then is centrifuged into three basic components: red blood cells, PRP and platelet-poor plasma. The PRP component is collected via manufactures recommendation, drawn into sterile syringes, and prepared for injection into the patient. 0.1cc of 10% CaCl2 per 1ml of PRP will be added and mixed into the PRP solution for injections on one side of the face.
  Injections will be completed using Softfil micro-cannulas inserted via a small puncture through the patients' skin to dissect into the subcutaneous plane

SUMMARY:
The purpose of the study is to determine the efficacy of platelet-rich plasma (PRP) as a cosmetic facial injectable filler to treat tear troughs deformities secondary to volume loss and skin laxity in the infra-orbital region. Patients will receive injections of PRP on the left side, and PRP with A VectraH1 3D camera will be used to quantify the volume of the infra-orbital region before treatment, at 1, 3, 6 and 12 months post treatment. The objective is to quantify the amount of volume gained in the region as well as to assess duration of volumization after PRP treatment and also if volumization results are permanent.

DETAILED DESCRIPTION:
The purpose of this study is to determine if PRP facial filler injections will provide effective long-term restoration of facial volume, specifically at the tear troughs. The study is a controlled trial. The attending surgeon and residents will perform the procedure. Pre-treatment photographs will be obtained of the patient using a VectraH1 3D head & neck camera. The provider will complete PRP injections first on the left side followed by PRP with calcium chloride on the right side. At no point during the study will we deviate from the standard of care for treatment with PRP or PRP with CaCl2. 0.1cc of 10% calcium chloride per 1mL of platelet rich plasma will be mixed. The volume of PRP and will be used upon the discretion of provider for treatment of the cosmetic facial deformity.

One of the most common filler materials used today are hyaluronic acid derivatives [13]. While these types of fillers offer certain advantages over bovine and collagen derived materials that may require skin testing prior to treatment; they can be expensive and will require ongoing injections as they absorb [14]. Autogenous fillers such as autogenous fat can offer a permanent solution, which may therefore decrease the net cost compared to hyaluronic acid derived fillers, but has higher morbidity associated with the fat harvesting and transfer [15-17]. PRP as a filler material may be the least expensive option with the lowest morbidity even if the effects are not yet proven to be permanent.

To evaluate whether the PRP facial filler treatment provides long term restoration of facial volume, patients will return for additional photographs and data collection using the VectraH1 3D head & neck camera at one, three, six and twelve months after treatment. The primary outcome will be the amount of facial volume achieved in the tear troughs, as assessed with the VectraH1 3D head & neck camera and VECTRA Capture Analysis module software to measure volume differences (cm3) pre- and post-treatment.

The Canfield VectraH1 3D head & neck camera is a high resolution device that captures the highest details and measures volume differences and contour changes of the face and neck. The camera allows for quantification of subsurface skin conditions using proprietary RBX® technology, allows for visualization of the degree of contour change with color distance mapping, allows for automated measurements to allow patients to understand their current conditions and visualize their post-treatment appearance. In contrast to previous 3D imaging systems, the VectraH1 is a low cost, highly portable system designed for facial imaging that has become very popular in cosmetic practice. It is a validated metric and is used within the cosmetic surgery community. The validation of tools used to measure surgical outcomes is fundamental for high-quality practice and outcomes research and studies performed with the VectraH1 show the system is accurate and comparable to other 3D imaging systems on the market such as 3dMDFace system. The advantage of the VectraH1 is the portability of the camera as opposed to a stationary system.

VectraH1 3D head & neck camera would be an asset for any training programs participating in cosmetic surgery and would be an asset to our study for several reasons. The 3D camera would allow us to most accurately assess the volume changes in the nasojugal folds using the color distance mapping technology to visualize the results rather than relying on sequential 2D imaging and clinical measurement, further reinforcing our study data and obtaining the most accurate results possible. Currently the VectraH1 3D head & neck camera is widely utilized in the cosmetic surgery community with testimonials from facial plastic surgeons warranting the ease of use of the product, the increase in patient satisfaction when using the camera as well as an exponential increase in use of facial fillers and fat transfer due to the realistic simulations the camera provides [18]. When patients can see the difference a filler procedure or fat transfer can provide prior to treatment, patient have a realistic expectation for what to expect and allow patients to see themselves as we do as cosmetic surgeons. This camera is a practice changer in that the clinician benefits with the most accurate imaging technology available for pre-treatment simulations and assessments as well as for the patient by offering the most realistic expectations for their individual treatment and opens the door for procedures they may not have previously considered. The use of this product would benefit our residency immensely in the cosmetic domain and keep us up-to-date with the technology that is available and utilized in private practice. This would also benefit the Air Force by opening the door for more potential candidates for cosmetic surgical procedures that may have foregone treatment once they can visualize the benefits of the procedures.

This study is projected to last approximately one year per patient. The tear trough facial volumes will be measured pre-procedure and at 1, 3, 6 and 12 months following the procedure. The data will be reviewed after an N of 50 is reached to assess the results. An interval evaluation of the data at N of 20 and 40 will be analyzed to evaluate for concerns regarding efficacy. The facial volumes reported will enable us to draw conclusions as to the overall success of the PRP facial filler injections with and without calcium chloride, and allow us to validate it's long term use as a viable facial filler.

At the conclusion of the study, the patient will have the option to treat the remaining tear trough with the PRP with calcium chloride facial filler treatment if results between the two sides are noticeable, unless if determined to be contraindicated by the attending physician.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* Patients with deepened tear troughs who are scheduled to receive PRP injections in DGMC Oral & Maxillofacial Surgery clinic.

Exclusion Criteria:

* Pregnant or nursing
* History of any type of neuralgia or paresthesia, or paresis
* Allergy or contraindication to lidocaine
* Use of hyaluronic acid in last 12 months
* Use of facial filler in last 12 months
* Have an active inflammatory or infectious process at the injection site
* Documented bleeding dyscrasias to include thrombocytopenia or anemia, platelet or clotting factor disorders
* Severe coronary artery disease
* No history of facial trauma
* No midface deformity or herniation of fat pads
* Active use of aspirin or anticoagulants
* History of keloids or hypertrophic scarring

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-01-31 (Estimated); Primary Completion 2019-02-01 (Estimated); Study Completion 2019-02-01 (Estimated)

PRIMARY OUTCOMES:
Facial volume changes | 1, 3, 6 and 12 months
  The study control will be the facial volumes recorded for each patient on both sides of the face prior to injections of PRP and PRP with CaCl2. These values will be obtained through analysis using the VectraH1 3D head & neck camera and recorded pre-operatively.

CONTACTS AND LOCATIONS:
Overall Officials: Ryan M Diepenbrock, DMD, Principal Investigator — David Grant Medical Center

IPD SHARING:
Plan to Share IPD: Yes
IPD will be available to other researches to include the efficacy of PRP and PRP with CaCl for use as a permanent facial filler if successful. Data shared will be sustainable volume measurements with PRP and PRP with CaCl.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: At the completion of the study to be completed in Q1 or Q2 of 2018.
Access Criteria: IPD Sharing Access Criteria not yet determined.

REFERENCES:
- [Background] Loesch MM, Somani AK, Kingsley MM, Travers JB, Spandau DF. Skin resurfacing procedures: new and emerging options. Clin Cosmet Investig Dermatol. 2014 Aug 28;7:231-41. doi: 10.2147/CCID.S50367. eCollection 2014. PMID 25210469
- [Background] Boxrud, C., et al., Infraorbital discoloration: Dark Circles-An Anatomic Analysis and Treatment. Plastic Surgery Key.
- [Background] Marx RE. Platelet-rich plasma: evidence to support its use. J Oral Maxillofac Surg. 2004 Apr;62(4):489-96. doi: 10.1016/j.joms.2003.12.003. No abstract available. PMID 15085519
- [Background] Rodriguez-Flores J, Palomar-Gallego MA, Enguita-Valls AB, Rodriguez-Peralto JL, Torres J. Influence of platelet-rich plasma on the histologic characteristics of the autologous fat graft to the upper lip of rabbits. Aesthetic Plast Surg. 2011 Aug;35(4):480-6. doi: 10.1007/s00266-010-9640-5. Epub 2010 Dec 24. PMID 21184066
- [Background] Li K, Li F, Li J, Wang H, Zheng X, Long J, Guo W, Tian W. Increased survival of human free fat grafts with varying densities of human adipose-derived stem cells and platelet-rich plasma. J Tissue Eng Regen Med. 2017 Jan;11(1):209-219. doi: 10.1002/term.1903. Epub 2014 Jun 30. PMID 24978937
- [Background] Hamilton B, Tol JL, Knez W, Chalabi H. Exercise and the platelet activator calcium chloride both influence the growth factor content of platelet-rich plasma (PRP): overlooked biochemical factors that could influence PRP treatment. Br J Sports Med. 2015 Jul;49(14):957-60. doi: 10.1136/bjsports-2012-091916. Epub 2013 Jun 15. PMID 23770705
- [Background] Smith, A., Procedure For Autologous Thrombin Activation of Platelets in Platelet Rich Plasma (PRP). Oral Health, 2006.
- [Background] Cervelli V, Nicoli F, Spallone D, Verardi S, Sorge R, Nicoli M, Balzani A. Treatment of traumatic scars using fat grafts mixed with platelet-rich plasma, and resurfacing of skin with the 1540 nm nonablative laser. Clin Exp Dermatol. 2012 Jan;37(1):55-61. doi: 10.1111/j.1365-2230.2011.04199.x. PMID 22182435
- [Background] Keller MW, Han PP, Galarneau MR, Gaball CW. Characteristics of maxillofacial injuries and safety of in-theater facial fracture repair in severe combat trauma. Mil Med. 2015 Mar;180(3):315-20. doi: 10.7205/MILMED-D-14-00345. PMID 25735023
- [Background] Cheng, X., et al., Preclinical Evaluation of Biomask Materials towards Facial Skin Regeneration. US Army Institute of Surgical Research (USAISR).
- [Background] Ayala, C., et al, Orbital Trauma and Nasoethmoid fractures. p. 289-314.
- [Background] Grahovac, T., et al., Interim Analysis of a Prospective Clinical Trial: Correlation of Biological Parameters with Clinical Outcome in Craniofacial Fat Grafting. Plastic Surgery Research Laboratory, McGowan Institute for Regenerative Medicine, University of Pittsburgh, PA.
- [Background] Kusin S, Lippitz J. Skin fillers. Dis Mon. 2009 Apr;55(4):236-56. doi: 10.1016/j.disamonth.2009.01.002. No abstract available. PMID 19286057
- [Background] Tran C, Carraux P, Micheels P, Kaya G, Salomon D. In vivo bio-integration of three hyaluronic acid fillers in human skin: a histological study. Dermatology. 2014;228(1):47-54. doi: 10.1159/000354384. Epub 2013 Dec 3. PMID 24503674
- [Background] Alijotas-Reig J, Fernandez-Figueras MT, Puig L. Inflammatory, immune-mediated adverse reactions related to soft tissue dermal fillers. Semin Arthritis Rheum. 2013 Oct;43(2):241-58. doi: 10.1016/j.semarthrit.2013.02.001. Epub 2013 May 2. PMID 23642806
- [Background] Eppley BL, Dadvand B. Injectable soft-tissue fillers: clinical overview. Plast Reconstr Surg. 2006 Sep 15;118(4):98e-106e. doi: 10.1097/01.prs.0000232436.91409.30. PMID 16980841
- [Background] Buck DW 2nd, Alam M, Kim JY. Injectable fillers for facial rejuvenation: a review. J Plast Reconstr Aesthet Surg. 2009 Jan;62(1):11-8. doi: 10.1016/j.bjps.2008.06.036. Epub 2008 Oct 31. PMID 18951862
- [Background] Liliana Camison, M., Michael Bykowski, MD, Wei Wei Lee, BS, Jesse A. Goldstein, MD, Joseph E. Losee, MD, Seth Weinberg, PhD, Validating Outcome Metrics: Accuracy of the VECTRA H1 Portable 3D Photogrammetry System for Facial Imaging Applications. 2016: University of Pittsburgh, Pittsburgh, PA, USA.